CLINICAL TRIAL: NCT00239356
Title: Aripiprazole (BMS-337039) for Outpatients With Schizophrenia Completing Aripiprazole Clinical Trials: A Non-Comparative Rollover Protocol
Brief Title: Aripiprazole for Schizophrenia Outpatients Completing BMS Clinical Trials
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN138-112
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AI (Experimental)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 10 - 30 mg, once daily, greater than 52 weeks depending upon Aripiprazole approval in respective country
  Other Names: Abilify; BMS-337039

SUMMARY:
The purpose of this study is to provide aripiprazole to schizophrenic outpatients and Community Treated Patients who are currently receiving aripiprazole therapy on another BMS sponsored clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving aripiprazole at time of screening
* Men and women ages 18 to 70

Exclusion Criteria:

* All patients previously discontinued from an aripiprazole study for any reason
* Active alcohol or substance abuse
* Patients who represent a significant risk of committing suicide
* Patients with clinically significant abnormal laboratory test results, vital signs or ECG findings

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2003-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- Canada (2):
  - Local Institution, Ottawa, Ontario
  - Local Institution, Sherbrooke, Quebec
- Croatia (2):
  - Local Institution, Rijeka
  - Local Institution, Zagreb
- Czechia (2):
  - Local Institution, Hradec Králové
  - Local Institution, Prague
- France (3):
  - Local Institution, Nantes Orvault
  - Local Institution, Rennes
  - Local Institution, Uzès
- Hungary (2):
  - Local Institution, Budapest
  - Local Institution, Győr
- Local Institution, Vught, Netherlands
- Poland (2):
  - Local Institution, Krakow
  - Local Institution, Poznan
- Local Institution, Bucharest, Romania
- Local Institution, Saint Petersburg, Russia
- South Africa (3):
  - Local Institution, Westdene, Free State
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Cape Town, Western Cape
- Local Institution, Antrim, Antrim, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study continued to provide aripiprazole post-study to schizophrenic and bipolar I disorder outpatients who had received aripiprazole on other Bristol-Myers Squibb Company (BMS)-sponsored clinical trials.
Pre-assignment Details: 119 enrolled, 117 treated. Reason(s) for not treated: 2 participants withdrew consent prior to treatment.
Groups:
- Aripiprazole 10 - 30 mg Once Daily (QD): Aripiprazole for schizophrenic participants: Tablets, Oral, 10 - 30 mg, once daily, greater than 52 weeks depending upon Aripiprazole approval in respective country.
- Aripiprazole 5 - 30 mg QD: Aripiprazole for Bipolar I Disorder participants: Tablets, Oral, 5 - 30 mg, once daily, greater than 52 weeks depending upon Aripiprazole approval in respective country.
Period: Overall Study
Arm/Group | Aripiprazole 10 - 30 mg Once Daily (QD) | Aripiprazole 5 - 30 mg QD
Started | 97 | 20
Completed | 58 | 11
Not Completed | 39 | 9
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 6 | 0
Not completed — Withdrawal by Subject | 15 | 6
Not completed — Lost to Follow-up | 3 | 0
Not completed — poor/non-compliance | 2 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Administrative reason | 0 | 1
Not completed — Drug available on market | 11 | 2

BASELINE CHARACTERISTICS:
Population: All treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole 10 - 30 mg Once Daily (QD) | Aripiprazole 5 - 30 mg QD | Total
Number analyzed (Participants) | 97 | 20 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (11.66) | 40.3 (11.78) | 39.5 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 2 | 37
  Male | 62 | 18 | 80
Region of Enrollment [Number; unit: participants]
  France | 24 | 0 | 24
  Hungary | 10 | 0 | 10
  Czech Republic | 3 | 0 | 3
  Canada | 11 | 0 | 11
  Poland | 7 | 0 | 7
  Romania | 4 | 0 | 4
  Croatia | 11 | 0 | 11
  Russian Federation | 9 | 0 | 9
  South Africa | 8 | 0 | 8
  Netherlands | 1 | 0 | 1
  United Kingdom | 2 | 0 | 2
  Germany | 2 | 0 | 2
  India | 0 | 20 | 20
  Israel | 1 | 0 | 1
  Spain | 3 | 0 | 3
  Switzerland | 1 | 0 | 1
Clinical Global Impression (CGI) Severity [Mean (Standard Deviation); unit: Units on a scale] — Clinical Global Impression (CGI) Severity Scores are measured on a scale of 1 to 7, with 1 being least severe and 7 being the most severe.
  Units on a scale | 2.6 (0.97) | 1.0 (0.00) | 2.3 (1.06)

OUTCOME MEASURES:

1. Primary Outcome: Mean Clinical Global Impression Severity Score (CGI-S) From Baseline Through End of Study- - Safety Population.
Description: Baseline is Day 1 of the study, prior to first dose. CGI-S is a questionnaire completed by the clinician which evaluates the severity of mental illness of a participant at a specific point in time. It consists of 7 categories with the lower categories indicating less illness and the higher numbered categories indicating greater severity of illness: 0=not assessed; 1=normal, not at all ill; 2=borderline mentally ill; 3= mildly ill; 4=moderately ill; 5= markedly ill; 6=severely ill; 7=among the most extremely ill.
Time Frame: Baseline to Week 348
Population: Safety Population - all participants who received at least one dose of drug. N=number of participants who were analyzed at each specific time point. Baseline N=97, 20 for first and second arms, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole 10 - 30 mg Once Daily (QD) | Aripiprazole 5 - 30 mg QD
Number analyzed (Participants) | 97 | 20
units on a scale
  Baseline | 2.6 (0.97) | 1.0 (0.00)
  Week 52 (N=67, 15) | 2.3 (0.75) | 1.1 (0.35)
  Week 108 (N=46,15) | 2.3 (0.66) | 1.1 (0.35)
  Week 156 (N=26,12) | 2.4 (0.80) | 1.1 (0.29)
  Week 212 (N=21,0) | 2.1 (0.96) | NA (NA) — All participants had dropped out or completed study in the Bipolar Disorder arm.
  Week 260 (N=8,0) | 1.9 (1.13) | NA (NA) — All participants had dropped out or completed study in the Bipolar Disorder arm.
  Week 316 (N=5,0) | 2.4 (1.14) | NA (NA) — All participants had dropped out or completed study in the Bipolar Disorder arm.
  Week 348 (N=5,0) | 2.4 (1.14) | NA (NA) — All participants had dropped out or completed study in the Bipolar Disorder arm.

2. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Adverse Events (AEs), and Discontinuation Due to an AE - Safety Population
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: Baseline to Week 348
Population: Safety Population: all participants with at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Aripiprazole 10 - 30 mg Once Daily (QD) | Aripiprazole 5 - 30 mg QD
Number analyzed (Participants) | 97 | 20
participants
  Death | 0 | 0
  Serious Adverse Events | 13 | 0
  Adverse Events | 47 | 14
  Discontinuations due to AEs | 6 | 0

3. Secondary Outcome: Mean Exposure to Aripiprazole at Days 541 to 630, Days 721 to 810 and Days 1081 to 1170 - Safety Population
Description: Mean exposure is mean number of milligrams per day (mg/day) of aripiprazole administered to the participants.
Time Frame: Day 1 to Day 1170
Population: N=number of participants receiving drug at Days indicated.
Measure: Mean (Full Range); unit: mg/day
Arm/Group | Aripiprazole 10 - 30 mg Once Daily (QD) | Aripiprazole 5 - 30 mg QD
Number analyzed (Participants) | 97 | 20
mg/day
  Days 541 to 630 (N=57, 17) | 20.25 [10.0 to 30.0] | 13.53 [10.0 to 30.0]
  Days 721 to 810 (N=44, 15) | 20.55 [10.0 to 30.0] | 13.67 [10.0 to 30.0]
  Days 1081 to 1170 (N=27, 12) | 23.20 [10.0 to 60.0] | 14.7 [10.0 to 30.0]

4. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Chemistry Laboratory Abnormalities During Treatment - Safety Population
Description: Clinically relevant abnormalities: greater than, equal to (>=); less than, equal to (<=). Upper limits of normal (ULN). milligram per deciliter (mg/dL); milliequivalent per liter (mEq/L); nanograms per milliliter (ng/mL);outside of normal range inclusive (): alanine transaminase (ALT>= 3*ULN; aspartate aminotransferase (AST >=3*ULN; alkaline phosphatase >=3*ULN; total bilirubin >= 2.0 mg/dL; blood urea nitrogen >= 30mg/dL; calcium (8.40 - 9.90 mg/dL); chloride (85.00 - 108.00 mEq/L); total cholesterol (140.0 - 200.0 mg/dL); cholesterol high density (HDL) and low density (LDL) lipoprotein (39.0 - 116.0 mg/dL); creatine kinase (15.0 - 170.0 U/L); creatinine >=2.0 mg/dL; prolactin (3.00 - 29.00 ng/mL); sodium (136.0 - 144.0 mEq/L); Glucose fasting (70.0 - 110.0 mg/dL); triglycerides (58.0 - 164.0 mg/dL; uric acid male >= 10.5, female >= 8.5mg/dL. Baseline is Day 1 of the study, prior to study drug administration.
Time Frame: Baseline to end of study (Week 348)
Population: Safety Population: all participants with at least 1 dose of study drug. Number of participant analyzed is given as N in each category of laboratory test.
Measure: Number; unit: participants
Arm/Group | Aripiprazole 10 - 30 mg Once Daily (QD) | Aripiprazole 5 - 30 mg QD
Number analyzed (Participants) | 97 | 20
participants
  Total Bilirubin (N=78, 18) | 4 | 0
  Blood urea nitrogen (N=37, 18) | 1 | 0
  Total Calcium (N=76, 18) | 1 | 0
  Serum chloride (N=62, 17) | 1 | 0
  Cholesterol HDL Fasting (N=44, 13) | 17 | 9
  Cholesterol LDL Fasting (N=47, 13) | 13 | 0
  Total Cholesterol Fasting (N=55, 16) | 15 | 0
  Creatine Kinase (N=64, 18) | 2 | 0
  Creatinine (N=81, 18) | 1 | 0
  Glucose, Fasting serum (N=61, 15) | 12 | 8
  Glucose, serum (N=37, 2) | 2 | 0
  Prolactin (N=63, 18) | 8 | 1
  Sodium, serum (N=76, 17) | 1 | 0
  Triglycerides Fasting (N=59, 16) | 17 | 2
  Uric Acid (N=71, 17) | 1 | 0

5. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Hematology Laboratory Abnormalities During Treatment - Safety Population
Description: Clinically relevant laboratory abnormality: Hemoglobin male <= 11.5 g/dL; female <= 9.5 g/dL. Hematocrit male <= 37 and 3 point decrease from baseline (BL); female <=32 and 3 point decrease from BL. Leukocytes <= 2800 mm^3 or >= 16000 mm^3; eosinophils >=10%. Baseline is Day 1 of the study, prior to study drug administration.
Time Frame: Baseline to end of study (Week 348)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Aripiprazole 10 - 30 mg Once Daily (QD) | Aripiprazole 5 - 30 mg QD
Number analyzed (Participants) | 97 | 20
participants
  Eosinophils, relative (N=80, 18) | 1 | 3
  Hematocrit (N=80, 16) | 1 | 1
  Hemoglobin (N=81, 18) | 2 | 1
  Leukocytes (N=81, 18) | 1 | 1

6. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Vital Sign Abnormality During Treatment - Safety Population
Description: Vital signs include standing, sitting and supine systolic and diastolic blood pressure, measured in millimeters of mercury (mmHg) and standing, sitting and supine heart rate, measured in beats per minute. Baseline (BL) is Day 1 of the study, prior to study drug administration. Criteria for identifying vital sign values as clinically relevant: Systolic blood pressure (criterion value=90-180 mmHg) change relative to baseline: increase of greater than, equal to (>=) 20; decrease of >= 20 mmHg. Diastolic blood pressure (criterion value=50 - 105 mmHg) change relative to baseline: increase of >= 15; decrease of >= 15 mmHg. Heart rate (criterion value=50-120bpm) change relative to baseline: increase >=15; decreased >= 15 mmHg. To be clinically significantly abnormal: value must meet the criterion value and also represent a change from the participant's pre-treatment value of at least the magnitude shown in the change relative to baseline.
Time Frame: Baseline to end of study (Week 348)
Population: Safety Population: all participants with at least 1 dose of study drug. Number of participants analyzed is given as N in each vital sign parameter and includes those treated participants with vital sign measurements.
Measure: Number; unit: participants
Arm/Group | Aripiprazole 10 - 30 mg Once Daily (QD) | Aripiprazole 5 - 30 mg QD
Number analyzed (Participants) | 97 | 20
participants
  Standing Systolic decrease (N=87,18) | 3 | 0
  Standing Diastolic increase (N=87,18) | 1 | 0
  Supine Diastolic increase (N=79,20) | 1 | 0
  Sitting Diastolic increase (N=61,5) | 2 | 0
  Standing Heart Rate increase (N=87,18) | 3 | 0
  Orthostatic Hypotension (N=78, 18) | 1 | 0

7. Secondary Outcome: Number of Participants With Potentially Clinically Relevant ECG Abnormalities During Treatment - Safety Population
Description: Potentially clinically relevant abnormality or change relative to baseline: sinus tachycardia: >= 120 beats per minute (bpm) and increased >= 15 bpm; sinus bradycardia: <= 50 bpm and decrease >= 15 bpm; supraventricular tachycardia, ventricular tachycardia, atrial fibrillation, atrial flutter: not present to present. First degree atrioventricular (A-V) block: PR interval(beginner of P wave to beginning of complex of Q, R, and S waves) >= 0.20 seconds (sec) and increase >= 0.05 sec; second and third degree A-V block, right bundle branch block (RBB) block, left bundle branch block (LBB) block: not present to present; other intraventricular block: QRS (complex of Q, R and S waves) >= 0.12 sec and increase >= 0.02 sec. Myocardial ischemia not present to present. QT interval with Bazett's correction (QTcB) or Fridericia's correction (QTcF) >= 450 milliseconds (msec) and elevation of 10% over baseline.
Time Frame: Baseline to end of study (Week 348
Population: Safety Population: all participants with at least 1 dose of study drug. Number of participants analyzed is given as N in each ECG parameter and includes those treated participants with ECG measurements.
Measure: Number; unit: participants
Arm/Group | Aripiprazole 10 - 30 mg Once Daily (QD) | Aripiprazole 5 - 30 mg QD
Number analyzed (Participants) | 97 | 20
participants
  Tachycardia (N=85, 16) | 0 | 1
  Bradycardia (N=85, 16) | 1 | 1
  Sinus Tachycardia (N=85, 16) | 0 | 1
  Sinus Bradycardia (N=85, 16) | 1 | 1
  First degree A-V Block (N=85, 16) | 10 | 0
  RBB Block (N=85, 16) | 1 | 0
  Pre-excitation syndrome (N=85, 16) | 1 | 0
  Other intraventricular Block (N=85, 16) | 7 | 2
  Myocardial Ischemia (N=85, 16) | 1 | 0
  QTcB (N=83, 16) | 11 | 4
  QTcF (N=83, 16) | 6 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected up to the participant's last visit. SAEs that occurred within 4 weeks after study discontinuation were included.
Description: Participants were to continue to receive study drug until: treatment intolerance, voluntary withdrawal, death, lost to follow up, no longer receiving benefit, the study drug was otherwise available through marketed means, the development of the study drug was terminated by the sponsor, or until 01 November 2012, whichever came first.
Groups:
- Bipolar I Disorder 5 - 30 mg QD: Aripiprazole for Bipolar I Disorder participants: Tablets, Oral, 5 - 30 mg, once daily, greater than 52 weeks depending upon Aripiprazole approval in respective country.
- Schizophrenia 10 - 30 mg QD: Aripiprazole for schizophrenic participants: Tablets, Oral, 10 - 30 mg, once daily, greater than 52 weeks depending upon Aripiprazole approval in respective country.
Arm/Group | Bipolar I Disorder 5 - 30 mg QD | Schizophrenia 10 - 30 mg QD
Serious Adverse Events (participants affected / at risk) | 0/20 | 13/97
Other Adverse Events (participants affected / at risk) | 10/20 | 22/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bipolar I Disorder 5 - 30 mg QD (N=20) | Schizophrenia 10 - 30 mg QD (N=97)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 2
Treatment noncompliance (Social circumstances) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Inadequate housing (Social circumstances) | 0 | 1
Psychosocial support (Surgical and medical procedures) | 0 | 4
Depression (Psychiatric disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bipolar I Disorder 5 - 30 mg QD (N=20) | Schizophrenia 10 - 30 mg QD (N=97)
Nasopharyngitis (Infections and infestations) | 3 | 4
Anxiety (Psychiatric disorders) | 0 | 6
Insomnia (Psychiatric disorders) | 1 | 5
Pyrexia (General disorders) | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Headache (Nervous system disorders) | 6 | 6
Vomiting (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.